CLINICAL TRIAL: NCT01127399
Title: Effects of Obesity on Airway Caliber and Airway Smooth Muscle Tone
Brief Title: Bariatric and Obstructive Lung Disease Study II
Acronym: BOLD II
Status: Terminated | Type: Observational
Why Stopped: Funding revoked
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NA_00027264; K23HL097081 (NIH)
Record Dates: First submitted 2010-05-19; First posted 2010-05-20 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Obesity; Asthma
MeSH Terms: conditions — Obesity; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Bariatric, nonasthma: Participants that will have had a bariatric surgery but do not have asthma.
- Bariatric, asthma: Participants that will have had a bariatric surgery and have been physician diagnosed with asthma prior to the surgery.
- Control, nonasthma: Healthy participants that who will not be getting a bariatric surgery and who do not have asthma.
- Control, asthma: Healthy participants that will not be having a bariatric surgery but do have asthma.

SUMMARY:
The prevalence of obesity and asthma has significantly increased over the past two decades. The purpose of this study is to try and understand the mechanism by which obesity leads to airway hyperresponsiveness (AHR), one of the defining features of asthma. This research is being done to determine how weight or body size affects airway size and airway smooth muscle (ASM) tone and function. The goal of the study will be to look at if and how, weight might affect lung functioning.

The investigators hypothesize that low lung volumes in obesity lead to AHR by reducing airway caliber causing increased ASM tone with impairment in deep inspiration (DI) response similar to what is seen in asthma.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* BMI over 35 kg/m2 (Bariatric) or BMI between 25 and 28 kg/m2 (Control)
* Physician diagnosis of asthma and on active asthma medication (if asthmatic)

Exclusion Criteria:

* Weight greater than 450 lbs
* Unstable cardiovascular disease
* Uncontrolled hypertension
* Renal failure on dialysis
* Cirrhosis
* Pregnant or lactating
* Bleeding disorders or Coumadin use
* Recent hospitalization for asthma in the past 3 months
* Active smoking or more than 10 pack year smoking history

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Bariatric Center at The Johns Hopkins University (Bariatric participants only), local community (Baltimore and Central Maryland area; control participants only)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle Clerisme-Beaty, MD, MHS, Principal Investigator — The Johns Hopkins University
Locations (1):
- The Johns Hopkins University, The Johns Hopkins Bayview Medical Campus, Baltimore, Maryland, United States